CLINICAL TRIAL: NCT04807959
Title: A Retrospective Study to Evaluate the Effectiveness of a Comprehensive Visceral Adiposity-Focused Anti-Obesity Program
Brief Title: Evaluation of the Effectiveness of a Comprehensive Visceral Adiposity-Focused Anti-Obesity Program
Status: Completed | Type: Observational
Sponsor: 20Lighter (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-443A
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Obesity, Morbid; Obesity, Visceral; Central Obesity; Metabolic Disease; Hypertension; Dyslipidemias; Type 2 Diabetes; Visceral Obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid; Obesity, Abdominal; Metabolic Diseases; Hypertension; Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 20Lighter Program Participants: All enrolled subjects will have completed a 20Lighter anti-obesity program prior to enrollment.
  Interventions: Other: 20Lighter anti-obesity program

INTERVENTIONS:
Other: 20Lighter anti-obesity program — A customized expert supervised 3-phase program including non-invasive proprietary nutritional, behavioral, and physiological components.

SUMMARY:
A retrospective review of body composition outcomes of participants of a comprehensive visceral-fat focused anti-obesity program. Data from approximately 2000-2500 participants are expected to be included in the study.

DETAILED DESCRIPTION:
This is a retrospective, multi-center clinical study to evaluate the efficacy of the 20Lighter comprehensive anti-obesity program in reducing body composition measures including body weight, body fat, visceral adiposity, intracellular fluid, and other metrics of interest. Anecdotal evidence on reductions of prescription medication, chronic health issues, and improvements in quality of life will be gauged via review of patient assessment forms and surveys.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25
* ability to stand on platform for body composition analysis

Exclusion Criteria:

* Pregnant at time of enrollment
* Breastfeeding at time of enrollment
* Undergoing treatment for cancer at time of enrollment
* History of major organ transplant with immunosuppressant medication
* Over the 70 years of age with diagnosis of three cardiovascular comorbidities at time of enrollment
* Adult with a vegetarian diet
* Diagnosis of psychiatric conditions including: schizophrenia, bipolar disorder, manic depression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 with overweight or obesity, and may have other comoribid conditions including hypertension, type 2 diabetes, dyslipidemia, cardiovascular disease (CVD), nonalcoholic fatty liver disease, sleep apnea, and other related health issues.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Reduction of Visceral Adiposity | Change from baseline to program completion (60 Days)
  % reduction of visceral adiposity (as measured by visceral fat rating) measured via an FDA-cleared Class 2 medical device with Bioelectrical Impedance Analysis (BIA) via bipolar foot electrodes.

SECONDARY OUTCOMES:
Reduction of Body Weight | Change from baseline to program completion (60 Days)
  % reduction of body weight measured via an FDA-cleared Class 2 medical device with Bioelectrical Impedance Analysis (BIA) via bipolar foot electrodes.
Reduction of Body Mass Index | Change from baseline to program completion (60 Days)
  % reduction of body mass index measured via an FDA-cleared Class 2 medical device with Bioelectrical Impedance Analysis (BIA) via bipolar foot electrodes.
Reduction of Body Fat | Change from baseline to program completion (60 Days)
  % reduction of body fat measured via an FDA-cleared Class 2 medical device with Bioelectrical Impedance Analysis (BIA) via bipolar foot electrodes.
Increase of Intracellular Fluid | Change from baseline to program completion (60 Days)
  % increase of intracellular fluid (as measured by body water %) measured via an FDA-cleared Class 2 medical device with Bioelectrical Impedance Analysis (BIA) via bipolar foot electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Barnes, PhD, Study Chair — 20Lighter

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Balasubramanian P, Longo VD. Growth factors, aging and age-related diseases. Growth Horm IGF Res. 2016 Jun;28:66-8. doi: 10.1016/j.ghir.2016.01.001. Epub 2016 Jan 7. PMID 26883276
- [Background] Barnosky AR, Hoddy KK, Unterman TG, Varady KA. Intermittent fasting vs daily calorie restriction for type 2 diabetes prevention: a review of human findings. Transl Res. 2014 Oct;164(4):302-11. doi: 10.1016/j.trsl.2014.05.013. Epub 2014 Jun 12. PMID 24993615
- [Background] Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Varady KA. Alternate day fasting and endurance exercise combine to reduce body weight and favorably alter plasma lipids in obese humans. Obesity (Silver Spring). 2013 Jul;21(7):1370-9. doi: 10.1002/oby.20353. Epub 2013 May 29. PMID 23408502
- [Background] Collier R. Intermittent fasting: the science of going without. CMAJ. 2013 Jun 11;185(9):E363-4. doi: 10.1503/cmaj.109-4451. Epub 2013 Apr 8. No abstract available. PMID 23569168
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- [Background] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Background] Eshghinia S, Mohammadzadeh F. The effects of modified alternate-day fasting diet on weight loss and CAD risk factors in overweight and obese women. J Diabetes Metab Disord. 2013 Jan 9;12(1):4. doi: 10.1186/2251-6581-12-4. PMID 23497604
- [Background] Hoddy KK, Kroeger CM, Trepanowski JF, Barnosky A, Bhutani S, Varady KA. Meal timing during alternate day fasting: Impact on body weight and cardiovascular disease risk in obese adults. Obesity (Silver Spring). 2014 Dec;22(12):2524-31. doi: 10.1002/oby.20909. Epub 2014 Sep 24. PMID 25251676
- [Background] Longo VD, Panda S. Fasting, Circadian Rhythms, and Time-Restricted Feeding in Healthy Lifespan. Cell Metab. 2016 Jun 14;23(6):1048-1059. doi: 10.1016/j.cmet.2016.06.001. PMID 27304506
- [Background] Mattson MP, Allison DB, Fontana L, Harvie M, Longo VD, Malaisse WJ, Mosley M, Notterpek L, Ravussin E, Scheer FA, Seyfried TN, Varady KA, Panda S. Meal frequency and timing in health and disease. Proc Natl Acad Sci U S A. 2014 Nov 25;111(47):16647-53. doi: 10.1073/pnas.1413965111. Epub 2014 Nov 17. PMID 25404320